CLINICAL TRIAL: NCT07251244
Title: Effects of a Nutritional Supplement and Functional Exercise Program on Seasonal Immunity, Perceived Health, and Oxidative Stress in Older Adults
Brief Title: Supplement and Exercise Effects on Stationary Immunity and Health in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan C. Colado, Professor of Physical Education, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-FIS-4026420
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Aging; Older Adults
Keywords: Older adults; Nutritional supplement; Functional exercise; Seasonal immunity; Oxidative stress; Multicomponent training; Healthy aging; Quality of life; Non-pharmacological intervention; Randomized controlled trial
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Exercise + nutritional supplement (EXNS) (Experimental): Participants in this group will receive an oral daily dose of the natural-origin nutritional supplement in combination with a supervised multicomponent functional exercise program (2 sessions per week, 45-60 minutes each) for 6 months.
  Interventions: Dietary Supplement: Group 1: Exercise + nutritional supplement (EXNS)
- Group 2: Exercise + placebo nutritional supplement (EXPlaNS) (Placebo Comparator): Participants in this group will receive a placebo supplement identical in appearance to the active supplement, together with the same multicomponent functional exercise program for 6 months.
  Interventions: Dietary Supplement: Group 2: Exercise + placebo nutritional supplement (EXPlaNS)

INTERVENTIONS:
Dietary Supplement: Group 1: Exercise + nutritional supplement (EXNS) — Participants in this group will receive an oral daily dose of the natural-origin nutritional supplement in combination with a supervised moderate-intensity multicomponent and functional exercise program (2 sessions per week, 45-60 minutes each) for 6 months, composed by three exercise blocks: 1) joint mobility and postural control exercises block, 2) explosive functional strength block with three sets of two strength exercises using elastic bands at 70% of 1RM and performed at maximum speed and, 3) coordination and agility exercises block.
  Arms: Group 1: Exercise + nutritional supplement (EXNS)
Dietary Supplement: Group 2: Exercise + placebo nutritional supplement (EXPlaNS) — Participants in this group will receive a placebo supplement identical in appearance to the active supplement, together with the same multicomponent functional exercise program for 6 months.
  Arms: Group 2: Exercise + placebo nutritional supplement (EXPlaNS)

SUMMARY:
The goal of this clinical trial is to learn whether a natural-origin nutritional supplement, combined with a moderate-intensity functional exercise program, can improve seasonal immunity, perceived health, and oxidative stress in older adults. The study will also assess the safety of this combined intervention.

The main questions it aims to answer are:

* Does the combination of supplementation and exercise enhance immune function during seasonal changes?
* Does it reduce oxidative stress and improve perceived health and functional capacity?

Researchers will compare a supplement to a placebo. All participants will follow the same supervised functional exercise program.

Participants will:

* Take a daily nutritional supplement for 6 months.
* Attend two weekly functional exercise sessions (60 minutes each), including mobility, explosive strength, and coordination/agility training.
* Complete three assessments (before, midway, and after the intervention) including blood tests, physical function evaluations, and quality of life questionnaires.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical trial with parallel groups, lasting a total of six months. Older adults (≥ 65 years) will participate and be randomly assigned to one of two intervention groups: nutritional supplement or placebo

All groups will follow a moderate-intensity multicomponent functional exercise program consisting of two weekly sessions of 60 minutes each, including mobility, explosive functional strength, and coordination/agility exercises. Three main assessments will be conducted (pre-, mid-, and post-intervention), during which blood samples will be collected to analyze immunological and oxidative stress biomarkers, along with data on functional, physiological, and quality of life variables.

The study is designed to evaluate the efficacy of combining nutritional supplementation with moderate physical exercise on seasonal immunity and overall health in older adults, ensuring blinding of both participants and investigators involved in data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older
* Functional independence, defined as the ability to perform activities of daily living without assistance
* Sufficient cognitive capacity to understand instructions and complete questionnaires, assessed through interview or brief cognitive screening if necessary
* Not immunosuppressed
* Not regular users of antioxidant or immunomodulatory supplements
* Ability and availability to attend exercise sessions and scheduled assessments throughout the six-month study period
* Commitment to maintain stable dietary and physical activity habits during the intervention

Exclusion Criteria:

* Active autoimmune diseases or clinically relevant immunosuppression
* Use of corticosteroids or immunosuppressive drugs in the 4 weeks prior to study initiation
* Active infection or compatible symptoms (fever, cough, diarrhea) in the 2 weeks prior to any measurement
* Unstable cardiovascular conditions or medical contraindications for moderate physical exercise
* Moderate to severe cognitive impairment that prevents proper participation in the scheduled activities
* Participation in another clinical trial in the last 3 months
* Known allergy or hypersensitivity to the supplement or any of its excipients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Changes in inteleukin 6 (IL-6) | Pre-, mid-, and post-intervention of 6 months
  Serum IL-6 levels will be collected through a blood sample in the morning in a fasted state to assess systemic inflammation and immunity
Changes in tumor necrosis factor alfa (TNF-α) | Pre-, mid-, and post-intervention of 6 months
  Serum TNF-α levels will be collected through a blood sample in the morning in a fasted state to assess chronic inflammation and immune state
Changes in immunoglobulin A and G (IgA, IgG) | Pre-, mid-, and post-intervention of 6 months
  IgA and IgG levels will be collected through a blood sample in the morning in a fasted state to assess immunological state.
Change in high-sensitivity C-reactive protein (hs-CRP) | Pre-, mid-, and post-intervention of 6 months
  Serum hs-CRP levels will be collected through a blood sample in the morning in a fasted state to assess systemic inflammatory state.
Complete blood count with leukocyte differential for neutrophil-to-lymphocyte ratio (NLR) calculation | Pre-, mid-, and post-intervention of 6 months
  Blood count with leukocyte levels will be collected through a blood sample in the morning in a fasted state to assess the NLR
Changes in interferon gamma (IFN-γ) | Pre-, mid-, and post-intervention of 6 months
  Serum IFN-γ levels will be collected through a blood sample in the morning in a fasted state to assess immunological and inflammatory state
Change in F2-isoprostanes | Pre-, mid-, and post-intervention of 6 months
  Serum F2-isoprostanes levels will be collected through a blood sample in the morning in a fasted state to assess the lipid peroxidation
Change in reduced glutathione (GSH) | Pre-, mid-, and post-intervention of 6 months
  Serum GSH levels will be collected through a blood sample in the morning in a fasted state to assess the thiol state/antioxidant response.
Change in total antioxidant capacity (TAC) | Pre-, mid-, and post-intervention of 6 months
  Serum TAC levels will be collected through a blood sample in the morning in a fasted state to assess the antioxidant response.

SECONDARY OUTCOMES:
Change in quality of life | Pre-, mid-, and post-intervention of 6 months
  Quality of life will be assessed through the WHOQOL-OLD tool
Change in general health perception | Pre-, mid-, and post-intervention of 6 months
  General health perception will be assessed through the EQ-5D-5L (EuroQol Group) tool
Change in gastrointestinal symptoms and gut health | Pre-, mid-, and post-intervention of 6 months
  Gastrointestinal symptoms and gut health will be assessed through the GSRS tool
Change in frequency and duration of minor illnesses | Pre-, mid-, and post-intervention of 6 months
  Frequency and duration of minor illnesses will be assessed through the Jackson Cold Scale.
Adherence to supplement and exercise | Every day for nutritional supplement and each exercise session during the 6 months of intervention.
  Adherence to supplement and exercise will be assessed through ad hoc questionnaire
Satisfaction with the intervention | Mid- and post-intervention of 6 months
  Satisfaction with the intervention will be assessed through ad hoc questionnaire
Change in distance covered/aerobic capacity | Pre-, mid-, and post-intervention of 6 months
  Distance covered/aerobic capacity will be assessed through the 6- Minute walking test
Changes in lower limb strength | Pre-, mid-, and post-intervention of 6 months
  Lower limb strength will be assessed through the 30-second Chair Stand Test
Changes in agility and dynamic balance | Pre-, mid-, and post-intervention of 6 months
  Agility and dynamic balance will be assessed through the Timed Up and Go Test
Changes in handgrip strength | Pre-, mid-, and post-intervention of 6 months
  Handgrip strength will be assessed through the Handgrip dynamometry (Jamar Hand Dynamometer).
Changes in resting heart rate and blood pressure | Pre-, mid-, and post-intervention of 6 months
  Resting heart rate and blood pressure will be assessed through a validated oscillometric sphygmomanometer
Changes in intraocular pressure | Pre-, mid-, and post-intervention of 6 months
  Intraocular pressure will be assessed through a non-contact tonometer
Changes in body composition | Pre-, mid-, and post-intervention of 6 months
  Whole body composition will be assessed through the Bioelectrical impedance analysis (Tanita BC-418). Total body mass, fat mass, lean mass and total body water mass will be measured.
Demographic characteristics | Pre-, mid-, and post-intervention of 6 months
  Age, sex, BMI, regular medication will be assessed.
Baseline physical activity level | Pre-, mid-, and post-intervention of 6 months
  Baseline physical activity level will be assessed through the IPAQ-short form questionnaire
Change in Frailty index | Pre-, mid-, and post-intervention of 6 months
  Frailty index will be assessed through the FRAIL Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Physical activity and Sport Science Faculty, Valencia, Valencia, Valencia, Valencia, Spain